CLINICAL TRIAL: NCT04331782
Title: Integration of Mental Health in HIV Clinic to Increase the Success of Antiretroviral Treatment: Screening for Depression Disorders in People With HIV in Hospitals
Brief Title: Integration of Mental Health in HIV Clinic to Increase the Success of ARV Treatment in PLWHA in Hospitals
Status: Completed | Type: Observational
Sponsor: Ina-Respond (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other)
Responsible Party: Sponsor
Other Study IDs: INA104.02
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: HIV/AIDS; Depression
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Integration of mental health in HIV clinics is needed in order to accelerate fast track 90-90-90 for controlling HIV. Symptoms of depression are sometimes difficult to recognize. In people living with HIV (PLWHA), depression that fails to be recognized and uncontrolled increases the risk of unsuccessful antiretroviral treatment and mortality.

The main purpose of this study is to estimate the proportion of depressive disorders in people living with HIV. The study included adult HIV patients aged ≥18 years, both men and women, who had received ARV treatment for at least six months, with no history of being diagnosed with depression.

DETAILED DESCRIPTION:
This study was a cross-sectional, non-intervention and multicenter in adults with HIV-AIDS (PLWHA) who were treated at a hospital who had received ARV treatment for at least six months, without a history of being diagnosed with depression.

Patients from HIV outpatient clinics in each research hospital were briefed on the study and offered to participate. Furthermore, based on the assessment of inclusion and exclusion criteria, PLWHA who meet the requirements were recruited and data were collected.

Sociodemographic data, HIV risk factors, risk behaviors, clinical characteristics such as duration of HIV, family history of mental illness, AIDS-related illnesses, other serious non-AIDS-related illnesses, treatment (antiretroviral (ARV) and non-ARV) and history ARV treatment response (HIV and CD4 viral load) were collected from each participant. In addition, a rapid screening for depressive disorders was carried out using the Patient Health Questionnaire-9 (PHQ-9) which was translated and validated in Indonesian. The PHQ-9 questionnaire was filled in by the patient with the assistance of health personnel. The total PHQ-9 questionnaire score were added up and the severity of depression associated with the score was reported to the patient's physician for further management.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years.
2. HIV positive based on diagnosis standards of care in research hospitals.
3. Have received ARV treatment for at least six months.
4. Without a history of being diagnosed with a depressive disorder beforehand.
5. Has been given an explanation before the research and give approval after the explanation.

Exclusion Criteria:

1. Being pregnant / nursing.
2. Currently undergoing a period of detention.
3. Being seriously ill (according to the doctor's justification at the hospital).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included adult HIV patients aged ≥18 years, both men and women, who had received ARV treatment for at least six months, with no history of being diagnosed with depression from HIV outpatient clinics in research hospital in Indonesia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of depressive disorders in PLWHA in hospitals. | [Time Frame: 3 months] [No Safety Issue]
  Number in percentage for Proportion of depressive disorders in PLWHA in hospitals.

SECONDARY OUTCOMES:
Distribution of the severity of depressive disorders in PLWHA | [Time Frame: 3 months] [No Safety Issue]
  Distribution of the severity of depressive disorders in PLWHA catagorized into minimal, mild, moderate, moderate-severe and severe
The correlation of depression with various factors. | [Time Frame: 3 months] [No Safety Issue]
  The correlation of depression with various factors: the Risk behavior in the past 30 days, socio-demographic, clinical characteristic and ARV response history.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Muhammad Karyana, MPH, Principal Investigator — National Institute of Health Research and Development, Ministry of Health Republic of Indonesia
Locations (4):
- Indonesia (4):
  - Site 600 : Adam Malik Hospital, Medan, North Sumatra
  - Site 650: Budi Kemuliaan Hospital, Batam, Riau Islands
  - Site 630: M. Ansari Saleh Hospital, Banjarmasin, South Kalimantan
  - Site 640: St. Carolus Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: No